CLINICAL TRIAL: NCT03868358
Title: Effect of Intermittent Theta Burst Stimulation (iTBS) for Alleviating Symptoms of Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WANG KAI (Other)
Responsible Party: Sponsor-Investigator, WANG KAI, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab Anhui Medical University, PRC, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ahmu-sjnk-scz
Record Dates: First submitted 2019-03-03; First posted 2019-03-11 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia; Functional Magnetic Resonance Imaging; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Stimulation (Active Comparator): Real Stimulation: active transcranial magnetic stimulation(Intermittent Theta Burst Stimulation).Participants will receive active TMS once daily for two weeks
  Interventions: Device: transcranial magnetic stimulation
- Sham Stimulation (Placebo Comparator): Sham Stimulation:no stimulation.Participants will receive sham TMS once daily for two weeks
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — The stimulations were performed by MagStim Rapid2. Participants in active comparator will receive active transcranial magnetic stimulation(Real Stimulation) daily for two weeks.
  Participants in sham comparator will receive no stimulation(Sham Stimulation) daily for two weeks

SUMMARY:
To investigate the treatment effect of intermittent theta-burst transcranial magnetic stimulation on symptomatic relief of schizophrenia patients, and the underlying neural mechanism by functional MRI and the resting electroencephalogram

DETAILED DESCRIPTION:
All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after intermittent theta-burst transcranial magnetic stimulation (iTBS) treatment. Patients were randomly allocated to iTBS group and the sham group by coin toss. There are about 30 patients in each group.The decision to enroll a patient was always made prior to randomization. Patients were studied using a double-blind design. Study participants, clinical raters, and all personnel responsible for the clinical care of the patient remained masked to allocated condition and allocation parameters. Only iTBS administrators had access to the randomization list; they had minimal contact with the patients, and no role in assessing the Positive and Negative Syndrome Scale (PANSS). Each patient would be treated for continuous 14 days by iTBS.Before the iTBS treatment, PANSS and Clinical Global Impression-severity of illness (CGI-SI) at baseline were obtained by a trained investigator to assess baseline severity of their symptoms. Scale for the Assessment of Negative Symptoms (SANS) and Scale for Assessment of Positive Symptoms (SAPS) were respectively supplemented to evaluate the severity of symptoms in different dimensions,.The patients had receiving a battery measure of neuropsychological tests (standardized tests to investigate their cognitive problems, anxiety and depressive symptoms in daily life), magnetic resonance imaging scan in multimodalities, electroencephalography (EEG), event-related potentials during stop signal test and Iowa-gambling test record. Other behavioral tests including intertemporal decision,spatial n-back test record.

After the last treatment, the Positive and Negative Syndrome Scale were obtained, as well as the Global Index of Safety to assess adverse events of the treatment. Patients were instructed to focus their answers on the past 14 days. The patients had also receiving a battery measure of neuropsychological tests, magnetic resonance imaging scan in multimodalities, and EEG record.Clinical Global Impression-global improvement (CGI-GI), Clinical Global Impression-efficacy index (CGI-EI) were evaluated at the end of treatment.

40-60 days after the last treatment, participants were interviewed to obtain the Positive and Negative Syndrome Scale,SAPS,SANS and HAMA,HAMD. They were instructed to focus their answers on the past week. Additionally, they were also asked to assess the battery of neuropsychological tests, and have magnetic resonance imaging scan in multimodalities, and EEG record. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Patients met diagnostic criteria for schizophrenia or schizoaffective disorder using the Structural Clinical Interview for Diagnostic and Statistical Manual Diploma in Social Medicine (DSM)-IV (SCID, Version 2.0).
* Patients remain their psychotropic medication at steady dosages for at least 4 weeks prior to study entry and for the duration of the trial.
* Verbal intelligence quotient > 85 as measured by using a Chinese version of the National Adult Reading Test.

Exclusion Criteria:

* History of significant head trauma or neurological disorders
* Alcohol or drug abuse Focal brain lesions on T1- or T2-weighted fluid-attenuated inversion-recovery magnetic resonance images
* a prior history of a seizure not induced by drug withdrawal,first degree relative with epilepsy, significant neurological illness or head trauma, endocrine disease, such as thyroid disease, significant unstable medical condition, recent aggression or other forms of behavioral dyscontrol
* left-handedness, pregnancy
* estimated intelligence quotient<80
* current alcohol or drug abuse
* inability to provide informed consent.
* Hamilton Anxiety Rating Scale or the Hamilton Depression Rating Scale score > 14

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-21 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Positive And Negative Syndrome Scale(PANSS) | Baseline and 2 weeks post-treatment,and follow-up
  The improvment in PANSS scores will constitute the major research outcome measure used to assess response to rTMS,reflecting the symptom improvment in patients

SECONDARY OUTCOMES:
Scale for the Assessment of Positive Symptoms (SAPS) | Baseline and 2 weeks post-treatment and follow-up
  The improvment in SAPS scores will constitute the major research outcome, and specifically reflect the degree of improvement in patients' positive symptoms
Scale for the Assessment of Negative Symptoms (SANS) | Baseline and 2 weeks post-treatment and follow-up
  The improvment in SANS scores will constitute the major research outcome, and specifically reflect the degree of improvement in patients' negative symptoms
Functional connectivity change of transcranial magnetic stimulation(iTBS and sham) | Baseline and 2 weeks post-treatment
  Functional MRI measures: the functional connectivity between stimulated target and the whole brain areas
EEG change of transcranial magnetic stimulation(iTBS and sham) | Baseline and 2 weeks post-treatment
  EEG measures: brain areas wave change of stimulation(iTBS and sham)
Intertemporal decision test | Baseline and 2 weeks post-treatment
  Intertemporal decision test is associated with the function of left dorsolateral prefrontal cortex
Spatial n-back test | Baseline and 2 weeks post-treatment
  Spatial n-back test will reflect the prefrontal function
Multidimensional Empathy Test | Baseline and 2 weeks post-treatment
  Multidimensional empathy Test is associated with the function of left dorsolateral prefrontal cortex

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China